CLINICAL TRIAL: NCT05804643
Title: Development and Optimization of Novel MRI Techniques on Evaluation of Therapeutic Effects for Lymphedema Secondary to Breast Cancer Treatment: An Integrated Study of Pre-clinical Animal Models and Clinical Follow-up
Brief Title: Novel MRI Techniques on Evaluation of Lymphedema
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 202301160RINA
Record Dates: First submitted 2023-03-08; First posted 2023-04-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Lymphedema of Upper Limb
Keywords: Lymphedema; supermicrosurgical technique; axillary procedures; pre-clinical animal model; diffusion MRI
MeSH Terms: conditions — Lymphedema | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer related lymphedema: Breast cancer related lymphedema cases receive observational magnetic resonance imaging before and after lymphovenous anastomosis.
  Interventions: Procedure: Diffusion magnetic resonance imaging

INTERVENTIONS:
Procedure: Diffusion magnetic resonance imaging — Free water elimination diffusion MRI and diffusion kurtosis MRI techniques

SUMMARY:
In this project, the investigators aim to investigate the imaging approaches for breast cancer-related secondary lymphedema. The clinical study aims to optimize the conventional MRI methods for mapping lymphedema and assess the post-surgical therapeutic effects in longitudinal follow-up studies. Additionally, a normal imaging database of lymphedema MRI images will be established for future reference. For pre-clinical animal study, investigators aim to develop and integrate two novel MRI methods, including free water elimination diffusion MRI and diffusion kurtosis MRI techniques. By integrating clinical and pre-clinical studies, the investigators aim to establish a precise imaging tool for evaluating the therapeutic effects of lymphedema for following translational applications.

DETAILED DESCRIPTION:
A total of three sub-projects will be conducted in this project. Sub-project 1 will establish a pre-clinical rat model for lymphedema and develop novel MRI methods, including diffusion kurtosis MRI and free water elimination diffusion MRI techniques, for mapping tissue characteristics of lymphedema. Sub-project 1 will be complemented with the clinical images provided by sub-project 2, yielding more information about the lymphedema. Sub-project 2 aims to optimize the clinical MRI methods for mapping lymphedema and quantitatively assess the severity of lymphedema. A normal imaging database will be established for reference. Sub-project 2 and sub-project 3 will be complementary in co-developing the image assessment of post-surgical therapeutic effect. Sub-project 3 will quantitatively evaluate the severity of lymphedema secondary to different kinds of axillary treatments by using the clinical MRI methods for establishing longitudinal monitoring and prediction approaches. It also focuses on the pre-surgical and post-surgical evaluation of lymphedema undergone supermicrosurgical technique by using the clinical MRI methods.

ELIGIBILITY:
Inclusion Criteria:

* adults with breast cancer related lymphedema

Exclusion Criteria:

* children younger than 20 years old
* pregnancy
* patients who have absolute contraindications regarding MRI scanning:

  1. The cardiac implantable electronic device (CIED) such as pacemakers, implantable cardioverter defibrillators (ICDs) and cardiac resynchronization therapy (CRT) devices.
  2. Metallic intraocular foreign bodies.
  3. Implantable neurostimulation systems
  4. Cochlear implants/ear implant: bone-anchored hearing aid (BAHA) cochlear implant type can be scanned on a 1.5-tesla scanner only after the patient removes the battery. Cochlear implant wrapping scheduling must take place before the patient's MRI appointment.
  5. Drug infusion pumps (insulin delivery, analgesic drugs, or chemotherapy pumps): If possible, the patient has to remove the device.
  6. Catheters with metallic components (Swan-Ganz catheter)
  7. Metallic fragments such as bullets, shotgun pellets, and metal shrapnel
  8. Cerebral artery aneurysm clips
  9. Magnetic dental implants
  10. Tissue expander
  11. Artificial limb
  12. Hearing aid

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with breast cancer related lymphedema
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline circumference of both arms at 3 months after lymphaticovenous anastomosis | baseline, 3 months after lymphaticovenous anastomosis
  circumference in cm
change from baseline volume of both arms at 3 months after lymphaticovenous anastomosis | baseline, 3 months after lymphaticovenous anastomosis
  volume in mL

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Kuo, Ph.D., Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- National Taiwan university hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fu MR. Breast cancer-related lymphedema: Symptoms, diagnosis, risk reduction, and management. World J Clin Oncol. 2014 Aug 10;5(3):241-7. doi: 10.5306/wjco.v5.i3.241. PMID 25114841
- [Background] Yang JC, Wu SC, Wang YM, Luo SD, Kuo SC, Chien PC, Tsai PY, Hsieh CH, Lin WC. Effect of Lymphaticovenous Anastomosis on Muscle Edema, Limb, and Subfascial Volume in Lower Limb Lymphedema: MRI Studies. J Am Coll Surg. 2022 Aug 1;235(2):227-239. doi: 10.1097/XCS.0000000000000236. Epub 2022 Apr 18. PMID 35839398
- [Background] Garza R 3rd, Skoracki R, Hock K, Povoski SP. A comprehensive overview on the surgical management of secondary lymphedema of the upper and lower extremities related to prior oncologic therapies. BMC Cancer. 2017 Jul 5;17(1):468. doi: 10.1186/s12885-017-3444-9. PMID 28679373
- [Background] Granzow JW, Soderberg JM, Kaji AH, Dauphine C. An effective system of surgical treatment of lymphedema. Ann Surg Oncol. 2014 Apr;21(4):1189-94. doi: 10.1245/s10434-014-3515-y. Epub 2014 Feb 13. PMID 24522988
- [Background] Winters H, Tielemans HJP, Hameeteman M, Paulus VAA, Beurskens CH, Slater NJ, Ulrich DJO. The efficacy of lymphaticovenular anastomosis in breast cancer-related lymphedema. Breast Cancer Res Treat. 2017 Sep;165(2):321-327. doi: 10.1007/s10549-017-4335-0. Epub 2017 Jun 12. PMID 28608029
- [Background] Executive Committee. The Diagnosis and Treatment of Peripheral Lymphedema: 2016 Consensus Document of the International Society of Lymphology. Lymphology. 2016 Dec;49(4):170-84. PMID 29908550
- [Background] Lohrmann C, Felmerer G, Foeldi E, Bartholoma JP, Langer M. MR lymphangiography for the assessment of the lymphatic system in patients undergoing microsurgical reconstructions of lymphatic vessels. Microvasc Res. 2008 May;76(1):42-5. doi: 10.1016/j.mvr.2008.03.003. Epub 2008 Mar 20. PMID 18456290
- [Background] Notohamiprodjo M, Weiss M, Baumeister RG, Sommer WH, Helck A, Crispin A, Reiser MF, Herrmann KA. MR lymphangiography at 3.0 T: correlation with lymphoscintigraphy. Radiology. 2012 Jul;264(1):78-87. doi: 10.1148/radiol.12110229. Epub 2012 Apr 20. PMID 22523325
- [Background] Franconeri A, Ballati F, Panzuto F, Raciti MV, Smedile A, Maggi A, Asteggiano C, Esposito M, Stoppa D, Lungarotti L, Bortolotto C, Giardini D, De Silvestri A, Calliada F. A proposal for a semiquantitative scoring system for lymphedema using Non-contrast Magnetic Resonance Lymphography (NMRL): Reproducibility among readers and correlation with clinical grading. Magn Reson Imaging. 2020 May;68:158-166. doi: 10.1016/j.mri.2020.02.004. Epub 2020 Feb 10. PMID 32057940
- [Background] Crescenzi R, Donahue PMC, Hartley KG, Desai AA, Scott AO, Braxton V, Mahany H, Lants SK, Donahue MJ. Lymphedema evaluation using noninvasive 3T MR lymphangiography. J Magn Reson Imaging. 2017 Nov;46(5):1349-1360. doi: 10.1002/jmri.25670. Epub 2017 Feb 28. PMID 28245075
- [Background] Arrive L, Derhy S, El Mouhadi S, Monnier-Cholley L, Menu Y, Becker C. Noncontrast Magnetic Resonance Lymphography. J Reconstr Microsurg. 2016 Jan;32(1):80-6. doi: 10.1055/s-0035-1549133. Epub 2015 Mar 31. PMID 25826439
- [Background] Lohrmann C, Foeldi E, Speck O, Langer M. High-resolution MR lymphangiography in patients with primary and secondary lymphedema. AJR Am J Roentgenol. 2006 Aug;187(2):556-61. doi: 10.2214/AJR.05.1750. PMID 16861563
- [Background] Bae JS, Yoo RE, Choi SH, Park SO, Chang H, Suh M, Cheon GJ. Evaluation of lymphedema in upper extremities by MR lymphangiography: Comparison with lymphoscintigraphy. Magn Reson Imaging. 2018 Jun;49:63-70. doi: 10.1016/j.mri.2017.12.024. Epub 2018 Jan 3. PMID 29306049
- [Background] Hagmann P, Jonasson L, Maeder P, Thiran JP, Wedeen VJ, Meuli R. Understanding diffusion MR imaging techniques: from scalar diffusion-weighted imaging to diffusion tensor imaging and beyond. Radiographics. 2006 Oct;26 Suppl 1:S205-23. doi: 10.1148/rg.26si065510. PMID 17050517
- [Background] Basser PJ, Mattiello J, LeBihan D. MR diffusion tensor spectroscopy and imaging. Biophys J. 1994 Jan;66(1):259-67. doi: 10.1016/S0006-3495(94)80775-1. PMID 8130344
- [Background] Jensen JH, Helpern JA, Ramani A, Lu H, Kaczynski K. Diffusional kurtosis imaging: the quantification of non-gaussian water diffusion by means of magnetic resonance imaging. Magn Reson Med. 2005 Jun;53(6):1432-40. doi: 10.1002/mrm.20508. PMID 15906300
- [Background] Jensen JH, Helpern JA. MRI quantification of non-Gaussian water diffusion by kurtosis analysis. NMR Biomed. 2010 Aug;23(7):698-710. doi: 10.1002/nbm.1518. PMID 20632416
- [Background] Chhetri A, Li X, Rispoli JV. Current and Emerging Magnetic Resonance-Based Techniques for Breast Cancer. Front Med (Lausanne). 2020 May 12;7:175. doi: 10.3389/fmed.2020.00175. eCollection 2020. PMID 32478083
- [Background] Tang L, Zhou XJ. Diffusion MRI of cancer: From low to high b-values. J Magn Reson Imaging. 2019 Jan;49(1):23-40. doi: 10.1002/jmri.26293. Epub 2018 Oct 12. PMID 30311988
- [Background] Li Z, Li X, Peng C, Dai W, Huang H, Li X, Xie C, Liang J. The Diagnostic Performance of Diffusion Kurtosis Imaging in the Characterization of Breast Tumors: A Meta-Analysis. Front Oncol. 2020 Oct 27;10:575272. doi: 10.3389/fonc.2020.575272. eCollection 2020. PMID 33194685
- [Background] Liu W, Wei C, Bai J, Gao X, Zhou L. Histogram analysis of diffusion kurtosis imaging in the differentiation of malignant from benign breast lesions. Eur J Radiol. 2019 Aug;117:156-163. doi: 10.1016/j.ejrad.2019.06.008. Epub 2019 Jun 17. PMID 31307642
- [Background] Rosenkrantz AB, Padhani AR, Chenevert TL, Koh DM, De Keyzer F, Taouli B, Le Bihan D. Body diffusion kurtosis imaging: Basic principles, applications, and considerations for clinical practice. J Magn Reson Imaging. 2015 Nov;42(5):1190-202. doi: 10.1002/jmri.24985. Epub 2015 Jun 26. PMID 26119267
- [Background] Collier Q, Veraart J, Jeurissen B, Vanhevel F, Pullens P, Parizel PM, den Dekker AJ, Sijbers J. Diffusion kurtosis imaging with free water elimination: A bayesian estimation approach. Magn Reson Med. 2018 Aug;80(2):802-813. doi: 10.1002/mrm.27075. Epub 2018 Feb 2. PMID 29393531
- [Background] Bergamino M, Walsh RR, Stokes AM. Free-water diffusion tensor imaging improves the accuracy and sensitivity of white matter analysis in Alzheimer's disease. Sci Rep. 2021 Mar 26;11(1):6990. doi: 10.1038/s41598-021-86505-7. PMID 33772083